CLINICAL TRIAL: NCT02001909
Title: Single-center, Open-label, Non-randomized, Two-period Sequential Treatment Study to Assess the Effect of Neomycin on the Pharmacokinetics of Regorafenib in Healthy Male Subjects
Brief Title: Effect of Neomycin on the Pharmacokinetics of Regorafenib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 16675; 2013-001721-18 (EudraCT Number)
Record Dates: First submitted 2013-11-28; First posted 2013-12-05 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Neoplasms
Keywords: Regorafenib; Neomycin; Cancer; Pharmacokinetics; Safety
MeSH Terms: conditions — Neoplasms | interventions — regorafenib; Neomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regorafenib (Experimental)
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)
- Neomycin (Experimental)
  Interventions: Drug: Neomycin

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — single oral dose (s.d.) 160 mg (four 40 mg tablets) of regorafenib on two occasions (Day 1, Period 1, and Day 1, Period 2) separated by a washout period of at least 14 days
  Arms: Regorafenib
Drug: Neomycin — 1 g tid (three times a day) regimen of Neomycin (oral) on five days in Period 2 starting 4 days before regorafenib intake on day 1 in period 2.
  Arms: Neomycin

SUMMARY:
To investigate the effect of neomycin on the pharmacokinetics (PK) of regorafenib in healthy male subjects

ELIGIBILITY:
Inclusion:

* Healthy male subjects
* Age: 18 to 45 years (inclusive) at the first screening examination/visit
* Body mass index (BMI): above/equal 18 and below 30 kg / m²
* Confirmation of the subject's health insurance coverage prior to the first screening examination/visit
* Subjects enrolled in this study must use adequate barrier birth control measures prior to, during the course of the study, and 3 months after the last administration of regorafenib. An adequate contraception includes the use of condoms or a vasectomy. In addition, adequate birth control measures for the subject's partner is required, such as a hormonal contraception with implants or combined oral contraceptives, certain intrauterine devices, bilateral tubal ligation, or hysterectomy.

Exclusion:

* Known or suspected hypersensitivity to regorafenib and/or neomycin
* Any illness or medical condition that is unstable or could jeopardize the safety of the subject and his compliance in the study
* Clinically significant illness within 30 days prior to Day 1, Period 1.
* Regular use of medicines at the time of screening, including herbal supplements and high dose vitamins
* Smoking; however, former smokers who have stopped smoking at least 3 months before the first study drug administration may be included
* Clinically relevant findings in the electrocardiogram (ECG)
* Clinically relevant findings in the complete physical examination
* Positive results for hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), human immune deficiency virus antibodies (anti-HIV 1+2) at screening.
* Positive urine drug screening

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
AUC (area under the plasma concentration vs. time curve) for regorafenib | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 and 192 hours post-dose
Cmax (maximum drug concentration) for regorafenib | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 and 192 hours post-dose

SECONDARY OUTCOMES:
AUC(0-24) (area under the plasma concentration vs. time curve) for regorafenib | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose
AUC(0-tlast) (area under the plasma concentration vs. time curve) for regorafenib | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 and 192 hours post-dose
AUC (area under the plasma concentration vs. time curve) for BAY75-7495 (M-2) and BAY81-8752 (M-5) | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 and 192 hours post-dose
Cmax (maximum drug concentration) for M-2 and M-5 | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 and 192 hours post-dose
tmax (time to reach maximum drug concentration in plasma after single dose) for regorafenib, M-2 and M-5 | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 and 192 hours post-dose
tlast (time of last concentration above lower limit of quantification) for regorafenib, M-2 and M-5 | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 and 192 hours post-dose
t1/2 (half-life associated with the terminal slope) for regorafenib, M-2 and M-5 | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 and 192 hours post-dose
AE,ur(0-72) (amount of drug excreted via urine during the collection interval 0-72 hours post administration) for metabolites BAY86-6651 (M-7) and BAY86-6652 (M-8) | 0-72 hours post dose
Number of participants with adverse events as a measure of safety and tolerability | Up to 30 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, State of Berlin, Germany

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/